CLINICAL TRIAL: NCT02532543
Title: Prospective, Comparative Volumetric Assessment of Alveolar Ridge Preservation Utilizing Different Bone Grafting Materials (SYMBIOS CORTICAL-CANCELLOUS GRANULE MIX; SYMBIOS OSTEOGRAF LD-300; OSTEOGRAF/N-300) Following Tooth Extraction
Brief Title: Comparative Volumetric Assessment of Alveolar Ridge Preservation Utilizing Different Bone Grafting Materials
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty in recruitment
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Dentsply International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-1114
Record Dates: First submitted 2015-08-21; First posted 2015-08-25 (Estimated); Results first posted 2019-12-09 (Actual); Last update posted 2019-12-09 (Actual); Status verified 2019-10

CONDITIONS: Tooth Fractures; Tooth Injuries; Tooth Diseases
MeSH Terms: conditions — Tooth Fractures; Tooth Injuries; Tooth Diseases | interventions — Transplantation, Homologous; Transplantation, Heterologous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group A- Allograft, Membrane (Active Comparator): Symbios mineralized cortical-cancellous granule mix, Symbios OsteoShield Collagen Resorbable Membrane
  Interventions: Biological: Allograft, Membrane
- Group B- Alloplast, Membrane (Active Comparator): Symbios OsteoGraf/LD-300, Symbios OsteoShield Collagen Resorbable Membrane
  Interventions: Biological: Alloplast, Membrane
- Group C- Xenograft, Membrane (Active Comparator): OsteoGraf/N-300 , Symbios OsteoShield Collagen Resorbable Membrane
  Interventions: Biological: Xenograft, Membrane
- Group D- Membrane (Active Comparator): Symbios OsteoShield Collagen Resorbable Membrane
  Interventions: Biological: Membrane

INTERVENTIONS:
Biological: Allograft, Membrane — Allograft, Membrane- Symbios mineralized cortical-cancellous granule mix, Symbios OsteoShield Collagen Resorbable Membrane
  Arms: Group A- Allograft, Membrane
Biological: Alloplast, Membrane — Alloplast, Membrane- Symbios OsteoGraf/LD-300, Symbios OsteoShield Collagen Resorbable Membrane
  Arms: Group B- Alloplast, Membrane
Biological: Xenograft, Membrane — Xenograft, Membrane- OsteoGraf/N-300,Symbios OsteoShield Collagen Resorbable Membrane
  Arms: Group C- Xenograft, Membrane
Biological: Membrane — Membrane - Symbios OsteoShield Collagen Resorbable Membrane
  Arms: Group D- Membrane

SUMMARY:
This study is intended to provide statistically robust evidence that Symbios Demineralized Cortical-cancellous granule mix, Symbios OsteoGraf LD-300, and OsteoGraf/N-300 combined with Symbios OsteoShield Collagen Resorbable Membrane can adequately support the alveolus during ridge augmentation procedures, reducing the dimensional changes of both the alveolus and the overlying soft tissues. Additionally, a comparison between each material will be made, providing further evidence of each materials' ability to preserve the alveolus. It is intended to define in objective terms the response of the hard and soft tissues to ridge augmentation.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent
2. ≥ 18 years and ≤ 75 years
3. Good physical health (ASAI/II)
4. Extraction of maxillary premolar, canine or incisor, or mandibular premolar and canine required
5. Teeth adjacent (mesial and distal) to study site must consist of two stable natural teeth with minimal restorations, without signs of periodontal bone loss (> 3 mm) and/or significant soft tissue deficiencies

Exclusion Criteria:

1. Buccal plate dehiscence and/or fenestration >3mm at study site following extraction
2. Untreated rampant caries and uncontrolled periodontal disease
3. Inadequate oral hygiene (estimated plaque score >20%)
4. Smokers using more than 10 cigarettes or equivalent per day
5. Smokeless tobacco use or e-cigarette use
6. Compromised physical health and/or uncontrolled or severe systemic diseases including:

   ASA III/IV Metabolic bone disease History of malignancy History or radiotherapy or chemotherapy for malignancy in the past 5 years History of autoimmune disease Long-term steroidal or antibiotic therapy Uncontrolled diabetes Known alcohol or drug abuse
7. Systemic or local disease or condition that would compromise post-operative healing
8. Use of any substance or medication that will influence bone metabolism
9. Known pregnancy
10. Unable or unwilling to return for follow-up visits for a period of 6 months
11. Unlikely to be able to comply with study procedures according to Investigators judgement
12. Involvement in the planning and conduct of the study
13. Previous enrollment or randomization of treatment in the present study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2018-02-12 (Actual); Study Completion 2018-02-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Reside, DDS MS, Principal Investigator — Dept. of Periodontology
Locations (1):
- University of North Carolina School of Dentistry, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schropp L, Wenzel A, Kostopoulos L, Karring T. Bone healing and soft tissue contour changes following single-tooth extraction: a clinical and radiographic 12-month prospective study. Int J Periodontics Restorative Dent. 2003 Aug;23(4):313-23. PMID 12956475
- [Background] Tan WL, Wong TL, Wong MC, Lang NP. A systematic review of post-extractional alveolar hard and soft tissue dimensional changes in humans. Clin Oral Implants Res. 2012 Feb;23 Suppl 5:1-21. doi: 10.1111/j.1600-0501.2011.02375.x. PMID 22211303
- [Background] Araujo MG, Lindhe J. Dimensional ridge alterations following tooth extraction. An experimental study in the dog. J Clin Periodontol. 2005 Feb;32(2):212-8. doi: 10.1111/j.1600-051X.2005.00642.x. PMID 15691354
- [Background] Ten Heggeler JM, Slot DE, Van der Weijden GA. Effect of socket preservation therapies following tooth extraction in non-molar regions in humans: a systematic review. Clin Oral Implants Res. 2011 Aug;22(8):779-88. doi: 10.1111/j.1600-0501.2010.02064.x. Epub 2010 Nov 22. PMID 21091540
- [Background] Darby I, Chen ST, Buser D. Ridge preservation techniques for implant therapy. Int J Oral Maxillofac Implants. 2009;24 Suppl:260-71. PMID 19885449
- [Background] Fienitz T, Schwarz F, Ritter L, Dreiseidler T, Becker J, Rothamel D. Accuracy of cone beam computed tomography in assessing peri-implant bone defect regeneration: a histologically controlled study in dogs. Clin Oral Implants Res. 2012 Jul;23(7):882-7. doi: 10.1111/j.1600-0501.2011.02232.x. Epub 2011 Jun 24. PMID 21707753
- [Background] Veyre-Goulet S, Fortin T, Thierry A. Accuracy of linear measurement provided by cone beam computed tomography to assess bone quantity in the posterior maxilla: a human cadaver study. Clin Implant Dent Relat Res. 2008 Dec;10(4):226-30. doi: 10.1111/j.1708-8208.2008.00083.x. Epub 2008 Apr 1. PMID 18384410
- [Background] Kim TS, Caruso JM, Christensen H, Torabinejad M. A comparison of cone-beam computed tomography and direct measurement in the examination of the mandibular canal and adjacent structures. J Endod. 2010 Jul;36(7):1191-4. doi: 10.1016/j.joen.2010.03.028. PMID 20630297
- [Background] Pertl L, Gashi-Cenkoglu B, Reichmann J, Jakse N, Pertl C. Preoperative assessment of the mandibular canal in implant surgery: comparison of rotational panoramic radiography (OPG), computed tomography (CT) and cone beam computed tomography (CBCT) for preoperative assessment in implant surgery. Eur J Oral Implantol. 2013 Spring;6(1):73-80. PMID 23513204
- [Background] Ganguly R, Ruprecht A, Vincent S, Hellstein J, Timmons S, Qian F. Accuracy of linear measurement in the Galileos cone beam computed tomography under simulated clinical conditions. Dentomaxillofac Radiol. 2011 Jul;40(5):299-305. doi: 10.1259/dmfr/72117593. PMID 21697155
- [Background] Tyndall DA, Price JB, Tetradis S, Ganz SD, Hildebolt C, Scarfe WC; American Academy of Oral and Maxillofacial Radiology. Position statement of the American Academy of Oral and Maxillofacial Radiology on selection criteria for the use of radiology in dental implantology with emphasis on cone beam computed tomography. Oral Surg Oral Med Oral Pathol Oral Radiol. 2012 Jun;113(6):817-26. doi: 10.1016/j.oooo.2012.03.005. PMID 22668710
- [Background] Watters W 3rd, Rethman MP, Hanson NB, Abt E, Anderson PA, Carroll KC, Futrell HC, Garvin K, Glenn SO, Hellstein J, Hewlett A, Kolessar D, Moucha C, O'Donnell RJ, O'Toole JE, Osmon DR, Evans RP, Rinella A, Steinberg MJ, Goldberg M, Ristic H, Boyer K, Sluka P, Martin WR 3rd, Cummins DS, Song S, Woznica A, Gross L; American Academy of Orthopedic Surgeons; American Dental Association. Prevention of Orthopaedic Implant Infection in Patients Undergoing Dental Procedures. J Am Acad Orthop Surg. 2013 Mar;21(3):180-9. doi: 10.5435/JAAOS-21-03-180. PMID 23457068
- [Background] Kurien S, Kattimani VS, Sriram RR, Sriram SK, Rao V K P, Bhupathi A, Bodduru RR, N Patil N. Management of pregnant patient in dentistry. J Int Oral Health. 2013 Feb;5(1):88-97. Epub 2013 Feb 26. PMID 24155583

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group A- Allograft, Membrane | Group B- Alloplast, Membrane | Group C- Xenograft, Membrane | Group D- Membrane
Started | 3 | 4 | 5 | 4
Completed | 3 | 4 | 4 | 4
Not Completed | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A- Allograft, Membrane | Group B- Alloplast, Membrane | Group C- Xenograft, Membrane | Group D- Membrane | Total
Number analyzed (Participants) | 3 | 4 | 5 | 4 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.3 (4.5) | 63.2 (5.7) | 49.2 (12.3) | 50.7 (20.7) | 53.0 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 3 | 2 | 6
  Male | 2 | 4 | 2 | 2 | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 4 | 5 | 4 | 16

OUTCOME MEASURES:

1. Primary Outcome: Total Mean Change in Bone Volume
Description: The change in bone volume at 3 months following extraction will be calculated using data from DICOM images acquired by Cone Beam Computed Tomography (CBCT) using 3D software
Time Frame: time of extraction to 3 months post extraction
Population: One participant was lost to follow up.
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | Group A- Allograft, Membrane | Group B- Alloplast, Membrane | Group C- Xenograft, Membrane | Group D- Membrane
Number analyzed (Participants) | 3 | 4 | 4 | 4
mm^3 | -91.64 (51.97) | -107.47 (52.31) | -77.31 (30.99) | -99.41 (66.00)
Statistical Analysis 1: Comparison: Group A- Allograft, Membrane vs Group B- Alloplast, Membrane vs Group C- Xenograft, Membrane vs Group D- Membrane; Test type: Superiority; p = 0.863, ANOVA

2. Secondary Outcome: Mean Osseous Dimensional Changes-Horizontal
Description: The amount of linear (mm) horizontal bone change at 3 months following tooth extraction at a position located 2mm and 4mm vertically away from the height of the buccal plate. Data will be calculated using data from DICOM images acquired by CBCT using 3D software.
Time Frame: time of extraction to 3 months post extraction
Population: One participant was lost to follow up. Measurements were taken at 2 and 4 mm instead of 3, 6 and 9 mm due to difficulties in data collection and patient variability
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Group A- Allograft, Membrane | Group B- Alloplast, Membrane | Group C- Xenograft, Membrane | Group D- Membrane
Number analyzed (Participants) | 3 | 4 | 4 | 4
mm
  2 mm from height of crest | -0.87 (0.98) | -1.30 (0.74) | -1.77 (0.42) | -1.62 (1.75)
  4 mm from height of crest | -1.03 (0.80) | -0.47 (0.57) | -0.92 (0.75) | -0.97 (1.48)
Statistical Analysis 1: Comparison: Group A- Allograft, Membrane vs Group B- Alloplast, Membrane vs Group C- Xenograft, Membrane vs Group D- Membrane; Comparison between each arm/group at 2 mm from the height of the bone crest; Test type: Superiority; p = 0.718, ANOVA
Statistical Analysis 2: Comparison: Group A- Allograft, Membrane vs Group B- Alloplast, Membrane vs Group C- Xenograft, Membrane vs Group D- Membrane; Comparison between each arm/group at 4 mm from the height of the bone crest; Test type: Superiority; p = 0.853, ANOVA

3. Secondary Outcome: Mean Osseous Dimensional Changes-Vertical
Description: The amount of linear (mm) vertical bone change at 3 months following tooth extraction at a position located mid-buccal, mid-palatal, mesial and distal of the extraction site. Data will be calculated using data from DICOM images acquired by CBCT using 3D software.
Time Frame: time of extraction to 3 months post extraction
Population: One participant was lost to follow up.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Group A- Allograft, Membrane | Group B- Alloplast, Membrane | Group C- Xenograft, Membrane | Group D- Membrane
Number analyzed (Participants) | 3 | 4 | 4 | 4
mm
  Mid Buccal | -1.23 (1.04) | -1.77 (1.58) | -2.00 (1.15) | -2.92 (3.14)
  Mid Palatal | -1.00 (0.40) | -1.02 (0.39) | -0.97 (0.46) | -1.02 (0.82)
  Mesial | -1.47 (0.55) | -0.87 (0.69) | -0.65 (1.14) | -1.60 (1.02)
  Distal | -1.07 (0.25) | -0.55 (0.46) | -0.60 (1.07) | -0.90 (0.62)
Statistical Analysis 1: Comparison: Group A- Allograft, Membrane vs Group B- Alloplast, Membrane vs Group C- Xenograft, Membrane vs Group D- Membrane; Comparison between each arm/group of change in mid buccal bone height; Test type: Superiority; p = 0.718, ANOVA
Statistical Analysis 2: Comparison: Group A- Allograft, Membrane vs Group B- Alloplast, Membrane vs Group C- Xenograft, Membrane vs Group D- Membrane; Comparison between each arm/group of change in mid palatal bone height; Test type: Superiority; p = 0.999, ANOVA
Statistical Analysis 3: Comparison: Group A- Allograft, Membrane vs Group B- Alloplast, Membrane vs Group C- Xenograft, Membrane vs Group D- Membrane; Comparison between each arm/group of change in mesial bone height; Test type: Superiority; p = 0.440, ANOVA
Statistical Analysis 4: Comparison: Group A- Allograft, Membrane vs Group B- Alloplast, Membrane vs Group C- Xenograft, Membrane vs Group D- Membrane; Comparison between each arm/group of change in distal bone height; Test type: Superiority; p = 0.729, ANOVA

4. Secondary Outcome: Total Mean Change in Soft Tissue Volume
Description: The change in soft tissue volume at 3 months following tooth extraction will be assessed through the use of 3D scans of patient dental models at two time points following extraction and ridge preservation at 3 months.
Time Frame: time of extraction to 3 months post extraction
Population: One participant was lost to follow up.
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | Group A- Allograft, Membrane | Group B- Alloplast, Membrane | Group C- Xenograft, Membrane | Group D- Membrane
Number analyzed (Participants) | 3 | 4 | 4 | 4
mm^3 | -99.44 (48.93) | -81.24 (13.24) | -82.71 (23.15) | -107.59 (38.59)
Statistical Analysis 1: Comparison: Group A- Allograft, Membrane vs Group B- Alloplast, Membrane vs Group C- Xenograft, Membrane vs Group D- Membrane; Test type: Superiority; p = 0.613, ANOVA

5. Secondary Outcome: Mean Soft Tissue Dimensional Changes-Horizontal
Description: The amount of linear (mm) horizontal soft tissue change at 3 months following tooth extraction at a position located 2mm and 4mm vertically away from the height of the buccal bone plate. Data will be calculated using data from DICOM images acquired by CBCT and overlaid 3D scans of patient dental models using 3D software.
Time Frame: time of extraction to 3 months post extraction
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Group A- Allograft, Membrane | Group B- Alloplast, Membrane | Group C- Xenograft, Membrane | Group D- Membrane
Number analyzed (Participants) | 3 | 4 | 4 | 4
mm
  2 mm from height of crest | -0.47 (0.47) | -0.67 (0.48) | -1.30 (0.82) | -0.87 (0.95)
  4 mm from height of crest | -0.40 (0.28) | -0.37 (0.25) | -0.70 (0.47) | -0.50 (1.14)
Statistical Analysis 1: Comparison: Group A- Allograft, Membrane vs Group B- Alloplast, Membrane vs Group C- Xenograft, Membrane vs Group D- Membrane; Comparison between each arm/group at 2 mm from the height of the bone crest; Test type: Superiority; p = 0.492, ANOVA
Statistical Analysis 2: Comparison: Group A- Allograft, Membrane vs Group B- Alloplast, Membrane vs Group C- Xenograft, Membrane vs Group D- Membrane; Comparison between each arm/group at 4 mm from the height of the bone crest; Test type: Superiority; p = 0.917, ANOVA

6. Secondary Outcome: Mean Soft Tissue Dimensional Changes-Vertical
Description: The amount of linear (mm) vertical soft tissue change at 3 months following tooth extraction at a position located mid-buccal, mid-palatal, mesial and distal of the extraction site. Data will be calculated using data from 3D scans of patient dental models using 3D software.
Time Frame: time of extraction to 3 months post extraction
Population: One participant was lost to follow up.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Group A- Allograft, Membrane | Group B- Alloplast, Membrane | Group C- Xenograft, Membrane | Group D- Membrane
Number analyzed (Participants) | 3 | 4 | 4 | 4
mm
  Mid Buccal | -1.60 (1.15) | -1.80 (0.62) | -1.72 (0.51) | -2.95 (1.75)
  Mid Palatal | -1.20 (0.36) | -1.00 (0.29) | -1.02 (0.68) | -1.30 (0.58)
  Mesial | -1.30 (1.04) | -1.02 (0.45) | -0.52 (0.59) | -1.37 (0.15)
  Distal | -1.53 (1.00) | -1.05 (0.66) | -1.12 (0.89) | -1.47 (0.32)
Statistical Analysis 1: Comparison: Group A- Allograft, Membrane vs Group B- Alloplast, Membrane vs Group C- Xenograft, Membrane vs Group D- Membrane; Comparison between each arm/group of change in mid buccal soft tissue height; Test type: Superiority; p = 0.353, ANOVA
Statistical Analysis 2: Comparison: Group A- Allograft, Membrane vs Group B- Alloplast, Membrane vs Group C- Xenograft, Membrane vs Group D- Membrane; Comparison between each arm/group of change in mid palatal soft tissue height; Test type: Superiority; p = 0.823, ANOVA
Statistical Analysis 3: Comparison: Group A- Allograft, Membrane vs Group B- Alloplast, Membrane vs Group C- Xenograft, Membrane vs Group D- Membrane; Comparison between each arm/group of change in mesial soft tissue height; Test type: Superiority; p = 0.243, ANOVA
Statistical Analysis 4: Comparison: Group A- Allograft, Membrane vs Group B- Alloplast, Membrane vs Group C- Xenograft, Membrane vs Group D- Membrane; Comparison between each arm/group of change in distal soft tissue height; Test type: Superiority; p = 0.756, ANOVA

7. Secondary Outcome: Soft Tissue Dimensional Change at Month 6
Description: The amount of soft tissue change will be assessed through the use of dental casts at two time points following extraction and ridge preservation at 6 months.
Time Frame: Month 6
Population: Data for the Month 6 timepoint was not collected
Arm/Group | Group A- Allograft, Membrane | Group B- Alloplast, Membrane | Group C- Xenograft, Membrane | Group D- Membrane
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From the signing of the Informed Consent form until study completion, a total of approximately 3 months
Arm/Group | Group A- Allograft, Membrane | Group B- Alloplast, Membrane | Group C- Xenograft, Membrane | Group D- Membrane
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/4 | 0/5 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/4 | 0/5 | 0/4
Other Adverse Events (participants affected / at risk) | 0/3 | 0/4 | 0/5 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-04): https://cdn.clinicaltrials.gov/large-docs/43/NCT02532543/Prot_SAP_000.pdf